CLINICAL TRIAL: NCT01694979
Title: Effect Of Variations In Forced Expiration Effort On Pelvic Floor Activation In Asymptomatic Women
Brief Title: Pelvic Floor Activity and Breathing in Women
Status: Completed | Type: Observational
Sponsor: Kitani, Lenore, PT (Other)
Responsible Party: Sponsor
Other Study IDs: L12-020
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Pelvic Floor; Respiration
Keywords: Pelvic floor; Rehabilitation; Respiration; Urinary incontinence
MeSH Terms: conditions — Respiratory Aspiration; Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: pelvic floor and breathing: This is a single group with repeated measures during variable breathing effort
  Interventions: Other: Minimum expiration effort; Other: Moderate expiration effort; Other: Maximum expiration effort

INTERVENTIONS:
Other: Minimum expiration effort — Subjects perform a forced expiration at minimum effort
Other: Moderate expiration effort — Subjects perform a forced expiration at moderate effort
Other: Maximum expiration effort — Subjects perform a forced expiration at maximum effort

SUMMARY:
The pelvic floor and diaphragm work together in many different functions. Two important functions are breathing and continence. The pelvic floor muscles have to lift and squeeze to maintain continence. Breathing, specifically breathing out, makes the pelvic floor lift. The investigators don't know how much the pelvic floor lifts and squeezes during different types of breathing out. The purpose of this study is to measure pelvic floor lift and squeeze during different types of breathing out.

DETAILED DESCRIPTION:
The pelvic floor (PF) activates automatically, both squeezing and lifting, during times of increased intra-abdominal pressure for postural stability and continence. Expiration additionally produces automatic activation of the PF. No study to date has investigated the effects of forced expiration on PF displacement and squeeze pressure. The purpose of this study was to investigate the effects of variations in forced expiration effort on PF muscles' automatic activation.

ELIGIBILITY:
Inclusion Criteria:

* women
* young (age 18-35)
* nulliparous
* pre-menopausal

Exclusion Criteria:

* pregnancy
* history of lower back or pelvic pain
* history of lower back or pelvic surgeries
* incontinence
* history of pelvic floor dysfunction
* diabetes
* endometriosis
* neuromuscular disease
* connective tissue disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Convenience sample from a University student, faculty and staff population.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenore J Kitani, B.S. PT, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Clinical Musculoskeletal Research Laboratory, Lubbock, Texas, United States

REFERENCES:
- [Background] Hodges PW, Sapsford R, Pengel LH. Postural and respiratory functions of the pelvic floor muscles. Neurourol Urodyn. 2007;26(3):362-71. doi: 10.1002/nau.20232. PMID 17304528
- [Background] Bo K, Berghmans B, Mørkved Siv, Van Kampen Marijke. Evidence-based physical therapy for the pelvic floor. 1st ed. Philedelphia, PA: Elsevier; 2007.
- [Background] Junginger B, Baessler K, Sapsford R, Hodges PW. Effect of abdominal and pelvic floor tasks on muscle activity, abdominal pressure and bladder neck. Int Urogynecol J. 2010 Jan;21(1):69-77. doi: 10.1007/s00192-009-0981-z. PMID 19730763
- [Background] Thompson JA, O'Sullivan PB. Levator plate movement during voluntary pelvic floor muscle contraction in subjects with incontinence and prolapse: a cross-sectional study and review. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Jun;14(2):84-8. doi: 10.1007/s00192-003-1036-5. Epub 2003 Apr 24. PMID 12851748
- [Background] Talasz H, Kremser C, Kofler M, Kalchschmid E, Lechleitner M, Rudisch A. Phase-locked parallel movement of diaphragm and pelvic floor during breathing and coughing-a dynamic MRI investigation in healthy females. Int Urogynecol J. 2011 Jan;22(1):61-8. doi: 10.1007/s00192-010-1240-z. Epub 2010 Aug 31. PMID 20809211
- [Background] Neumann P, Gill V. Pelvic floor and abdominal muscle interaction: EMG activity and intra-abdominal pressure. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(2):125-32. doi: 10.1007/s001920200027. PMID 12054180
- [Background] Smith MD, Coppieters MW, Hodges PW. Postural activity of the pelvic floor muscles is delayed during rapid arm movements in women with stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Aug;18(8):901-11. doi: 10.1007/s00192-006-0259-7. Epub 2006 Dec 1. PMID 17139463
- [Background] Ferreira CH, Barbosa PB, de Oliveira Souza F, Antonio FI, Franco MM, Bo K. Inter-rater reliability study of the modified Oxford Grading Scale and the Peritron manometer. Physiotherapy. 2011 Jun;97(2):132-8. doi: 10.1016/j.physio.2010.06.007. Epub 2010 Oct 22. PMID 21497247
- [Background] Frawley HC, Galea MP, Phillips BA, Sherburn M, Bo K. Reliability of pelvic floor muscle strength assessment using different test positions and tools. Neurourol Urodyn. 2006;25(3):236-242. doi: 10.1002/nau.20201. PMID 16299815
- [Background] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640
- [Background] Pregazzi R, Sartore A, Bortoli P, Grimaldi E, Troiano L, Guaschino S. Perineal ultrasound evaluation of urethral angle and bladder neck mobility in women with stress urinary incontinence. BJOG. 2002 Jul;109(7):821-7. doi: 10.1111/j.1471-0528.2002.01163.x. PMID 12135220
- [Background] Peschers UM, Gingelmaier A, Jundt K, Leib B, Dimpfl T. Evaluation of pelvic floor muscle strength using four different techniques. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(1):27-30. doi: 10.1007/s001920170090. PMID 11294527
- [Background] Thompson JA, O'Sullivan PB, Briffa K, Neumann P, Court S. Assessment of pelvic floor movement using transabdominal and transperineal ultrasound. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Jul-Aug;16(4):285-92. doi: 10.1007/s00192-005-1308-3. Epub 2005 Mar 22. PMID 15782286
- [Background] Shishido K, Peng Q, Jones R, Omata S, Constantinou CE. Influence of pelvic floor muscle contraction on the profile of vaginal closure pressure in continent and stress urinary incontinent women. J Urol. 2008 May;179(5):1917-22. doi: 10.1016/j.juro.2008.01.020. Epub 2008 Mar 18. PMID 18353401
- [Background] Bo K, Finckenhagen HB. Is there any difference in measurement of pelvic floor muscle strength in supine and standing position? Acta Obstet Gynecol Scand. 2003 Dec;82(12):1120-4. doi: 10.1046/j.1600-0412.2003.00240.x. PMID 14616257
- [Background] Constantinou CE, Hvistendahl G, Ryhammer A, Nagel LL, Djurhuus JC. Determining the displacement of the pelvic floor and pelvic organs during voluntary contractions using magnetic resonance imaging in younger and older women. BJU Int. 2002 Sep;90(4):408-14. doi: 10.1046/j.1464-410x.2002.02907.x. PMID 12175398
- [Background] Schaer GN, Koechli OR, Schuessler B, Haller U. Perineal ultrasound for evaluating the bladder neck in urinary stress incontinence. Obstet Gynecol. 1995 Feb;85(2):220-4. doi: 10.1016/0029-7844(94)00369-O. PMID 7824234
- [Background] Sapsford R. Rehabilitation of pelvic floor muscles utilizing trunk stabilization. Man Ther. 2004 Feb;9(1):3-12. doi: 10.1016/s1356-689x(03)00131-0. PMID 14723856
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Morin M, Bourbonnais D, Gravel D, Dumoulin C, Lemieux MC. Pelvic floor muscle function in continent and stress urinary incontinent women using dynamometric measurements. Neurourol Urodyn. 2004;23(7):668-74. doi: 10.1002/nau.20069. PMID 15382183
- [Background] Teleman PM, Gunnarsson M, Lidfeldt J, Nerbrand C, Samsioe G, Mattiasson A. Urethral pressure changes in response to squeeze: a population-based study in healthy and incontinent 53- to 63-year-old women. Am J Obstet Gynecol. 2003 Oct;189(4):1100-5. doi: 10.1067/s0002-9378(03)00539-8. PMID 14586362
- [Background] Bo K, Kvarstein B, Hagen RR, Larsen S. Pelvic floor muscle exercise for the treatment of female stress urinary incontinence: II. Validity of vaginal pressure measurements of pelvic floor muscle strength and the necessity of supplementary methods for control of correct contraction. Neurourol Urodyn 1990;9(5):479-487.
- [Background] Bo K, Constantinou C. Reflex contraction of pelvic floor muscles during cough cannot be measured with vaginal pressure devices. Neurourol Urodyn. 2011 Sep;30(7):1404. doi: 10.1002/nau.20993. Epub 2011 Mar 14. No abstract available. PMID 21404321
- [Background] Sherburn M, Bird M, Carey M, Bo K, Galea MP. Incontinence improves in older women after intensive pelvic floor muscle training: an assessor-blinded randomized controlled trial. Neurourol Urodyn. 2011 Mar;30(3):317-24. doi: 10.1002/nau.20968. Epub 2011 Jan 31. PMID 21284022
- [Background] Hung HC, Hsiao SM, Chih SY, Lin HH, Tsauo JY. An alternative intervention for urinary incontinence: retraining diaphragmatic, deep abdominal and pelvic floor muscle coordinated function. Man Ther. 2010 Jun;15(3):273-9. doi: 10.1016/j.math.2010.01.008. Epub 2010 Feb 24. PMID 20185357
- [Background] Dinc A, Kizilkaya Beji N, Yalcin O. Effect of pelvic floor muscle exercises in the treatment of urinary incontinence during pregnancy and the postpartum period. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1223-31. doi: 10.1007/s00192-009-0929-3. Epub 2009 Aug 1. PMID 19649552
- [Background] Miller JM, Perucchini D, Carchidi LT, DeLancey JO, Ashton-Miller J. Pelvic floor muscle contraction during a cough and decreased vesical neck mobility. Obstet Gynecol. 2001 Feb;97(2):255-60. doi: 10.1016/s0029-7844(00)01132-7. PMID 11165591
- [Background] Barbic M, Kralj B, Cor A. Compliance of the bladder neck supporting structures: importance of activity pattern of levator ani muscle and content of elastic fibers of endopelvic fascia. Neurourol Urodyn. 2003;22(4):269-76. doi: 10.1002/nau.10116. PMID 12808700